CLINICAL TRIAL: NCT06379113
Title: Gonadotropin-releasing Hormone Agonist (GnRHa) Plus Letrozole in Obese Progestin-insensitive Early-stage Endometrial Cancer Patients With Conservative Treatment
Brief Title: GnRHa + Letrozole in Obese Progestin-insensitive Endometrial Cancer Patients
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xiaojun Chen (Other)
Responsible Party: Sponsor-Investigator, Xiaojun Chen, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 53211030-2
Record Dates: First submitted 2024-02-21; First posted 2024-04-23 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Neoplasms; Atypical Endometrial Hyperplasia; Progesterone Resistance; Obesity
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia; Progesterone Resistance; Obesity | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Obese EEC group (Experimental): This group including 29 EEC cases. Interventional Study Model was Simon two-stage optimal design. Eleven patients were needed for the first stage, and if eight or more patients achieved CR at 28 weeks, the trial can enter into the second stage.
  Then every 12 to 16 weeks, an hysteroscope will be used to evaluate the endometrial condition, and the pathological findings will be recorded.
  Interventions: Drug: GnRH antagonist; Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: GnRH antagonist — Gonadotropin-releasing hormone analogue, intramuscular injection of 3.75mg will be given every 4 weeks, and the maximum treatment courses will be 6. If the patient get CR within 6 courses, another 2 courses will be used as consolidation therapy.
Drug: Letrozole 2.5mg — 2.5mg po qd.

SUMMARY:
To investigate the efficacy of GnRHa plus letrozole in obese progestin-insensitive EEC patients.

DETAILED DESCRIPTION:
There were more and more women with early endometrioid endometrial cancer (EEC) and atypical endometrial hyperplasia (EAH) who want to preserve fertility.

Approximately 70% to 80% of females who meet the criteria for conservation treatment are able to achieve CR after progestin therapy, with a median time of 6-7 months, but about 20% to 30% of patients get no response or need to take longer time to achieve remission (over one year). With long duration of treatment, there will be more side effects such as weight gain, impaired liver function, endometrial injury, ovarian reserve inhibition etc. which will decrease the efficacy of conservative treatment. Previous researches had shown that GnRHa plus letrozole could be a better second-line treatment for obese progestin-insensitive patients. Till now, no similar studies were found, so we design this study to explore the efficacy of GnRHa plus letrozole in obese progestin-insensitive EEC and EAH patients to provide new evidences for improving conservative treatment efficacy. We defined obese patients as these with BMI ≥ 30kg/m2.

This will be a single-centred prospective pilot study. Patients diagnosed as obese progestin-insensitive EEC by dilatation and curettage (D&C) or hysteroscopy will be enrolled. The primary endpoint is cumulative complete response (CR) rate at 28 weeks of treatment. The secondary endpoints include adverse events, duration of complete response, recurrent rate, pregnancy rate and quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed initial pathological diagnosis based upon hysteroscopy: histologically prove well-differentiated EEC G1 without myometrial invasion
* BMI≥30kg/m2
* No signs of suspicious extrauterine involvement on enhanced magnetic resonance imaging (MRI) or enhanced computed tomography (CT) or ultrasound
* Using progestin, any of the following therapy, as first-line treatment:

  1. Megestrol acetate ≥ 160 mg qd using, combined with Levonorgestrel Lntrauterine System (LNG-IUS) inserted or not
  2. Medroxyprogesterone acetate ≥ 250 mg qd using, combined with LNG-IUS inserted or not
  3. LNG-IUS inserted
* Progestin-insensitive:

  1. remained with stable disease after 7 months of progestin use
  2. did not achieve CR after 10 months of progestin use
* Have a desire for remaining reproductive function or uterus
* Good compliance with adjunctive treatment and follow-up

Exclusion Criteria:

* Combined with severe medical disease or severely impaired liver and kidney function
* Pathologically confirmed as endometrial cancer with suspicious myometrial invasion or extrauterine metastasis
* Patients with other types of endometrial cancer or other malignant tumors of the reproductive system
* Patients with breast cancer or other hormone- dependent tumors or diseases that cannot be used with GnRHa or Letrozole
* Strong request for uterine removal or other conservative treatment
* Known or suspected pregnancy
* Acute severe disease such as stroke or heart infarction or a history of thrombosis disease
* Smoker(>15 cigarettes a day)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rates within 28 weeks of treatment | Up to 28 weeks
  The cumulative 28-week CR rates will be calculated in two groups. Patients will be evaluated with an hysteroscopy every 12 to 16 weeks. For some may delay the evaluation as personal reasons, we define the primary outcome measure as complete response rates within 28 weeks of treatment.

SECONDARY OUTCOMES:
Adverse events | Through study completion, an average of 28 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be recorded, as well as incidence of adverse events.
Time to achieve complete response | Up to 28 weeks
  The median CR time will be calculated.
Relapse rates | Through study completion, an average of 2 years
Rates of fertility outcomes | Through study completion, an average of 2 years
Compliance | Through study completion, an average of 28 weeks
  Data on treatment and hysteroscopy management will be collected, and deviations from study protocol will be recorded in writing. For example, the time of drug interruptions due to related toxicities or AEs, and delay of hysteroscopy for personal reasons.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tenth People's Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Obstetrics and Gynecology Hospital, Fudan University, Shanghai

REFERENCES:
- [Background] Zhou S, Xu Z, Yang B, Guan J, Shan W, Shi Y, Chen X. Characteristics of progestin-insensitive early stage endometrial cancer and atypical hyperplasia patients receiving second-line fertility-sparing treatment. J Gynecol Oncol. 2021 Jul;32(4):e57. doi: 10.3802/jgo.2021.32.e57. PMID 34085795